CLINICAL TRIAL: NCT06086925
Title: A Window of Opportunity Study of Black Raspberry for Patients With Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: A Window of Opportunity Study of Black Raspberry for Patients With HNSCC
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study was not initiated due to funding constraints and will not proceed in its current design.
Sponsor: Mitchell Machtay (Other)
Responsible Party: Sponsor-Investigator, Mitchell Machtay, Professor of Radiation Oncology, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PSCI-21-223
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2024-07

CONDITIONS: Squamous Cell Carcinoma of the Oral Cavity or Oropharynx
Keywords: black raspberry; head and neck squamous cell carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: All subjects will be a part of the same treatment group and receive the same dosage.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BRB treatment (Experimental): Day 1 of BRB will be determined based upon the anticipated surgery day. Subjects will be instructed to consume a total dose of 5 Gm/day (orally) by taking one BRB five times a day: one upon waking in the morning, one in the morning, one at noon, one in the evening, and one at bedtime. BRB should not be given during meals and drinking. The subject should avoid eating for about 30 minutes before and after taking a BRB.
  Interventions: Drug: Black Raspberry

INTERVENTIONS:
Drug: Black Raspberry — Each BRB contains 1 gram of black raspberry powder equal to roughly 6 black raspberries.
  Other Names: BRB

SUMMARY:
The purpose of this phase 0 Window of Opportunity study is to have subjects with Head and Neck Squamous Cell Carcinoma (HNSCC) receive same dosage of Black Raspberry Extract between their cancer diagnosis and standard treatment (surgery). Tumor biopsies and research blood before and after the investigational treatment (Black Raspberry Extract lozenges) are collected for translational research. The investigational treatment is kept short to avoid delaying standard treatment.

DETAILED DESCRIPTION:
The global incidence of head and neck squamous cell carcinoma (HNSCC) currently rests at roughly 630,000 cases per year, with approximately half of all cases resulting in death. In the United States alone, an estimated 3% of all cancers diagnosed yearly are comprised of oral cavity and pharynx cancers, accounting for 63,000 cases per year and 13,000 related deaths. The high rates of incidence and prevalence in HNSCC are largely due to a lack of effective long term treatment. Treating cancer, including HNSCC at late stages even with recent advances in targeted therapies continues to be a major challenge and thus mechanistically-based effective strategies to manage and control this disease are urgently needed. Epidermal Growth Factor Receptor (EGFR) is over expressed in about 90% of HNSCC; it is associated with a poor prognosis and it is an attractive therapeutic target for HNSCC.

Many cultures throughout history and across the world have used plants and herbs to treat medical problems and a percentage of modern medicines have been extracted from plants.Black Raspberries (BRB), also referred to as "blackcaps", are an entirely natural resource available over-the-counter for purchase. BRB contains high concentrations of anthocyanins which serve as antioxidants that help prevent free radical damage in the body. Rich in levels of Vitamin A and calcium, these berries have not shown any adverse reaction upon consumption nor pose any threat when taken in conjunction with other medications. Researchers confirmed that 14-day before surgical administration of BRB troches significantly reduced the gene expression of many biomarkers that are consistently overexpressed in Oral Squamous Cell Carcinoma (OSCC).

The investigator proposes the possibility of introducing BRB that may improve biomarkers such as tumor suppressor p120ctn and reduce resistance modulated by EGFR and its pathways, and anticipates that the results of this clinical trial will not only demonstrate the highly safe and feasible nature of adding BRB to standard therapy, but that there will be considerable, favorable changes in the molecular biology of these patients' cancers and their immune status.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 18 years of age
2. Histology and/or pathology of untreated squamous cell carcinoma (SCC) of the oral cavity or oropharynx, greater than stage 0 and planned for definitive surgery
3. The cancer may be HPV+ or HPV-, as defined by biomarker testing such as p16 immunohistochemistry.
4. ECOG performance status 0-2
5. Confirmation of adequate tissue from previous biopsy for immunohistochemistry analysis
6. A surgery date must be anticipated to occur within 16 to 30 days after the first dose of BRB

Exclusion Criteria:

1. Inability to provide informed consent 2. Pregnancy or breast feeding 3. Chemotherapy with the exception of low dose chemo being used for non-cancer treatments (eg. methotrexate for rheumatoid arthritis etc.) 4. Known hypersensitivity to BRB

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
H-score complied through tumor analysis | From the start of the BRB through surgery, the average duration ranges from 16 to 30 days
  H-score is a quantitative variable and can be obtained from analyzing the tissue samples

SECONDARY OUTCOMES:
safety data collection | 7-10 days after BRB treatment to 21- 42 days after surgery
  All the adverse events will be summarized via frequency tables by type, grade, severity, and relationship to the study medicine

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Machtay, MD, Principal Investigator — Penn State Cancer Institute